CLINICAL TRIAL: NCT01927562
Title: Evaluation of the Fractyl Duodenal Remodeling System for the Treatment of Type 2 Diabetes
Brief Title: Initial Clinical Evaluation of an Endoscopic Therapy for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fractyl Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-10000
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Duodenal Treatment (Experimental): The Duodenal Remodeling procedure utilizes both a trans-oral over the wire and endoscopic approach to minimally invasively ablating and remodeling the duodenum.
  Interventions: Device: Fractyl Duodenal Remodeling System

INTERVENTIONS:
Device: Fractyl Duodenal Remodeling System

SUMMARY:
The purpose of this study is to assess the safety and feasibility of the Fractyl Duodenal Remodeling System for the treatment of patients with poorly controlled Type 2 Diabetes.

DETAILED DESCRIPTION:
The purpose of this protocol is to evaluate the initial safety profile of the Fractyl System and its effect on participants with Type 2 Diabetes. This will be determined through the monitoring of adverse events and outcome measures including Mixed Meal Tolerance Test (MMTT).

ELIGIBILITY:
Inclusion Criteria:

1. Participants Age > 28 years and ≤ 75 years
2. Male or Female
3. Participants with Type 2 Diabetes who are treated for ≤ 10 years and are on stable oral diabetic medications for a minimum of 3 months
4. Participants with an HbA1c > 7.5 and ≤ 10.0%
5. Participants with a BMI > 24 and < 40
6. Participants willing to comply with study requirements and able to understand and comply with informed consent
7. Participants who have signed an informed consent form

Exclusion Criteria:

1. Participants diagnosed with Type I Diabetes or with a history of ketoacidosis
2. Participants using insulin for more than 12 months
3. Participants with probable insulin production failure (defined as fasting C Peptide serum <1ng/mL)
4. Participants that have known autoimmune disease as evidenced by a positive anti glutamic acid decarboxylase (GAD) blood test
5. Participants requiring prescription anticoagulation therapy and/or dual anti-platelet therapy including aspirin who cannot discontinue their medication for 14 days before and 14 days after the procedure
6. Participants with iron deficiency anemia - either currently or in their history
7. Participants with current symptomatic hypocalcemia or vitamin D deficiency (routine calcium and/or vitamin D supplementation would not be excluded)
8. Participants with or a history of abnormalities of the GI tract preventing endoscopic access to the duodenum,
9. Participants with symptomatic gallstones or kidney stones at the time of screening
10. Participants with a history of pancreatitis
11. Participants with an active systemic infection
12. Participants with or a history of coagulopathy, upper gastro-intestinal bleeding c conditions such as ulcers, gastric varices, strictures, congenital or acquired intestinal telangiectasia
13. Participants with celiac disease
14. Participants with active malignancy. Those who have had remedial treatment and/or are cancer free for 5 years can be enrolled
15. Participants with known active hepatitis or active liver disease
16. Participants emotionally unstable or who exhibit psychological characteristics which, in the opinion of the Investigator, make the participant a poor candidate for clinical trial participation
17. Participants with previous GI surgery that could affect the ability to treat the duodenum such as participants who have had a Bilroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions
18. Participants unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during treatment through 2 weeks post procedure phase
19. Participants receiving weight loss medications such as Meridia, Xenical, or over the counter weight loss medications
20. Participant with a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
21. Participants with active and uncontrolled gastroesophageal reflux disease (GERD) defined as grade II esophagitis or greater
22. Participants with active illicit substance abuse or alcoholism
23. Participants participating in another ongoing investigational clinical trial
24. Participants taking corticosteroids or drugs known to affect GI motility (i.e. Reglan)
25. Participants who are not potential candidates for duodenal exclusion surgery or general anesthesia

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-07-13 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard R Gomez, MD, Principal Investigator — Centro Clinico De La Obesidad
Locations (1):
- INDISA, Santiago, Chile

REFERENCES:
- [Derived] Rajagopalan H, Cherrington AD, Thompson CC, Kaplan LM, Rubino F, Mingrone G, Becerra P, Rodriguez P, Vignolo P, Caplan J, Rodriguez L, Galvao Neto MP. Endoscopic Duodenal Mucosal Resurfacing for the Treatment of Type 2 Diabetes: 6-Month Interim Analysis From the First-in-Human Proof-of-Concept Study. Diabetes Care. 2016 Dec;39(12):2254-2261. doi: 10.2337/dc16-0383. Epub 2016 Aug 12. PMID 27519448

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A screening endoscopy is performed to visually examine the participant's GI tract to ensure they meet the requirements of the exclusion criteria concerning anatomical anomalies that would preclude the ability to complete the treatment. A biopsy is also taken to evaluate the baseline tissue.
Groups:
- Duodenal Treatment: Fractyl Duodenal Remodeling System
Period: Overall Study
Arm/Group | Duodenal Treatment
Started | 57
Completed | 19 (5 at M24, 2 at M30,12 at M36 due to two protocol changes moving followups from M24 to M30 to M36)
Not Completed | 38
Not completed — Lost to Follow-up | 30
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Duodenal Treatment
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Chile | 57

OUTCOME MEASURES:

1. Primary Outcome: Changed in Mixed Meal Tolerance From Baseline to 3 Months
Description: Improvement in fasting plasma glucose based on Mixed Meal Tolerance Test between baseline and 3 months
Time Frame: 3 months
Population: The 5 subjects who did not receive an ablation were excluded from the efficacy population, yielding 52 subjects in the efficacy population (as-treated population).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Duodenal Treatment
Number analyzed (Participants) | 52
mg/dL
  FPG with MMTT at 3 months | 145.3 (53.7)
  FPG with MMTT at Baseline | 180.9 (53.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from the time of informed consent through end of study (up to 36 months after study procedure).
Arm/Group | Duodenal Treatment
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 3/57
Other Adverse Events (participants affected / at risk) | 43/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duodenal Treatment (N=57)
procedural complication (Injury, poisoning and procedural complications) | 1 (1)
duodenal stenosis (Gastrointestinal disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duodenal Treatment (N=57)
abdominal distension (Gastrointestinal disorders) | 11 (12)
abdominal pain (Gastrointestinal disorders) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Change of bowel habit (Gastrointestinal disorders) | 4 (4)
dyspepsia (Gastrointestinal disorders) | 4 (4)
duodenal stenosis (Gastrointestinal disorders) | 3 (3)
duodenitis (Gastrointestinal disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 2 (2)
gastritis erosive (Gastrointestinal disorders) | 2 (2)
oesophagitis (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)
abdominal discomfort (Gastrointestinal disorders) | 1 (1)
abdominal pain lower (Gastrointestinal disorders) | 1 (1)
dental caries (Gastrointestinal disorders) | 1 (1)
dental discomfort (Gastrointestinal disorders) | 1 (1)
flatulence (Gastrointestinal disorders) | 1 (1)
gastric ulcer (Gastrointestinal disorders) | 1 (1)
gingival oedema (Gastrointestinal disorders) | 1 (1)
irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
regurgitation (Gastrointestinal disorders) | 1 (1)
polydipsia (Metabolism and nutrition disorders) | 9 (11)
hypoglycaemia (Metabolism and nutrition disorders) | 3 (3)
hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
gout (Metabolism and nutrition disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
nasopharyngitis (Infections and infestations) | 4 (4)
genital candidiasis (Infections and infestations) | 3 (3)
candida infection (Infections and infestations) | 1 (1)
gastroenteritis viral (Infections and infestations) | 1 (1)
influenza (Infections and infestations) | 1 (1)
rash pustular (Infections and infestations) | 1 (1)
tooth abcess (Infections and infestations) | 1 (1)
tooth infection (Infections and infestations) | 1 (1)
vulvovaginitis (Infections and infestations) | 1 (1)
depressed mood (Psychiatric disorders) | 3 (3)
depression (Psychiatric disorders) | 3 (3)
anxiety (Psychiatric disorders) | 2 (2)
stress (Psychiatric disorders) | 2 (2)
emotional distress (Psychiatric disorders) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1)
panic attack (Psychiatric disorders) | 1 (1)
polyuria (Renal and urinary disorders) | 9 (10)
renal colic (Renal and urinary disorders) | 2 (2)
nocturia (Renal and urinary disorders) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2)
contusion (Injury, poisoning and procedural complications) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
laceration (Injury, poisoning and procedural complications) | 1 (1)
meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
procedural headache (Injury, poisoning and procedural complications) | 1 (1)
procedural hypertension (Injury, poisoning and procedural complications) | 1 (1)
skin injury (Injury, poisoning and procedural complications) | 1 (1)
headache (Nervous system disorders) | 2 (2)
paraesthesia (Nervous system disorders) | 2 (2)
ageusia (Nervous system disorders) | 1 (1)
facial paresis (Nervous system disorders) | 1 (1)
neuropathy peripheral (Nervous system disorders) | 1 (1)
sensory loss (Nervous system disorders) | 1 (1)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
visual acuity reduced (Eye disorders) | 3 (3)
vision blurred (Eye disorders) | 2 (2)
retinopathy (Eye disorders) | 1 (1)
Acanthosis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
hypothyroidism (Endocrine disorders) | 2 (2)
lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
angina pectoris (Cardiac disorders) | 1 (1)
jaundice (Hepatobiliary disorders) | 1 (1)
heart rate decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information received by PRINCIPAL INVESTIGATOR from SPONSOR, including, but not limited to, the Protocol, and all information developed during the Study is confidential information ("Confidential Information"), which is the sole and exclusive property of SPONSOR during the period of this Agreement and subsequent thereto.

DOCUMENTS (2):
  • Study Protocol (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT01927562/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT01927562/SAP_000.pdf